CLINICAL TRIAL: NCT02483663
Title: Brain Regulation of Appetite in Twins
Acronym: BRAT
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Ellen Schur, MD, MS, Associate Professor, Medicine, University of Washington
Other Study IDs: 38970
Record Dates: First submitted 2015-06-17; First posted 2015-06-29 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Appetite
Keywords: Twins; Obesity; Appetite
MeSH Terms: conditions — Obesity | interventions — Magnetic Resonance Imaging; Absorptiometry, Photon; Surveys and Questionnaires; Drug Implants

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 27 Monozygotic Pairs
  Interventions: Device: Functional Magnetic Resonance Imaging; Radiation: Dual Energy X-ray absorptiometry; Other: Questionnaires; Other: Mood and Appetite Ratings; Other: Test Meals; Other: Computer Tests; Procedure: Intravenous Catheter (IV) placement
- 27 Dizygotic Pairs
  Interventions: Device: Functional Magnetic Resonance Imaging; Radiation: Dual Energy X-ray absorptiometry; Other: Questionnaires; Other: Mood and Appetite Ratings; Other: Test Meals; Other: Computer Tests; Procedure: Intravenous Catheter (IV) placement

INTERVENTIONS:
Device: Functional Magnetic Resonance Imaging — Measure brain activity.
  Other Names: fMRI
Radiation: Dual Energy X-ray absorptiometry — Body composition measurements.
  Other Names: DXA
Other: Questionnaires — Questionnaires related to: health, weight, sleep, mood, dietary habits, attitudes towards eating, how you describe yourself.
Other: Mood and Appetite Ratings — Answer questions about how you are feeling at the moment.
Other: Test Meals — Breakfast, a snack, and lunch provided during study visit.
Other: Computer Tests — Perform a series of computer tests to determine reaction time.
Procedure: Intravenous Catheter (IV) placement — Blood samples collected throughout regular intervals during the study visit day to measure levels of hormones involved in regulating appetite and body weight. We will also determine if twins are fraternal or identical and will examine DNA to see if participants carry two genes that affect appetite or body weight, the FTO gene and the MC4R gene.

SUMMARY:
Scientists are examining the genetic and environmental influences on appetite and weight gain. The main purpose of this study is to look at how genetic and environmental factors may influence how the brain regulates appetite and food intake. Understanding how the brain regulates appetite and food intake may eventually lead to new ways to help people avoid obesity or lose weight.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to come with their twin to the University of Washington (Seattle)
* Additional Criteria for Aim 1 random sample only: Member of randomly selected MZ pair or
* Additional criteria for Aim 2 random sample only: One member of MZ or same-sex DZ pair with BMI of at least 30 kg/m^2
* Additional criteria for Aim 3 sample only: Member of randomly selected MZ pair, and not BMI discordant ≥ 5 kg/m^2

Exclusion Criteria:

* History of weight loss surgery or active participation in weight loss program
* Major medical problem (e.g., diabetes, cancer)
* Current use of weight loss medications or other medications known to alter appetite
* Pregnancy or menopause
* MRI contraindication (i.e., implanted metal, claustrophobia)
* Lifetime eating disorder
* Current smoking
* Current heavy alcohol use (≥2 drinks per day for females and ≥ 3 drinks per day for males)
* Self-reported weight >330 pounds at time of phone screening. MRI cannot accommodate all shapes or weights. Inability to have MRI does not exclude subject from participating in other study procedures.
* BMI < 18.5 or > 45 kg/m^2
* Allergies to study foods or inability to taste
* Twins were raised apart
* Co-twin not eligible or not willing to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Monozygotic and dizygotic twins recruited from the University of Washington Twin Registry
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2010-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Meal-induced nutrient and hormonal changes in plasma (insulin, GLP-1, ghrelin, glucose) | Baseline
Brain activation during fMRI in satiety-related regions | Baseline
Body composition: fasting leptin and dual energy X-ray absorptiometry (DXA) | Baseline
DNA evaluation of FTO genotypes | Baseline
Objective satiety: caloric and macronutrient intake | Baseline
Subjective satiety: visual analog scale (VAS) scores and appeal ratings | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Schur, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Melhorn SJ, Askren MK, Chung WK, Kratz M, Bosch TA, Tyagi V, Webb MF, De Leon MRB, Grabowski TJ, Leibel RL, Schur EA. FTO genotype impacts food intake and corticolimbic activation. Am J Clin Nutr. 2018 Feb 1;107(2):145-154. doi: 10.1093/ajcn/nqx029. PMID 29529147
- [Derived] Mestre ZL, Melhorn SJ, Askren MK, Tyagi V, Gatenby C, Young L, Mehta S, Webb MF, Grabowski TJ, Schur EA. Effects of Anxiety on Caloric Intake and Satiety-Related Brain Activation in Women and Men. Psychosom Med. 2016 May;78(4):454-64. doi: 10.1097/PSY.0000000000000299. PMID 26867073
- [Derived] Melhorn SJ, Mehta S, Kratz M, Tyagi V, Webb MF, Noonan CJ, Buchwald DS, Goldberg J, Maravilla KR, Grabowski TJ, Schur EA. Brain regulation of appetite in twins. Am J Clin Nutr. 2016 Feb;103(2):314-22. doi: 10.3945/ajcn.115.121095. Epub 2016 Jan 6. PMID 26739033
- See also: UW Twin Registry — http://uwtwinregistry.org/